CLINICAL TRIAL: NCT05398471
Title: Observational Clinical Trial Appraising Medical Trial Experiences of Rheumatoid Arthritis Patients Participating In Clinical Research
Brief Title: Medical Trial: Appraising Medical Trial Experiences of Rheumatoid Arthritis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 58103638
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Historically, participation in clinical trials has been highly skewed towards specific demographic groups. However, research identifying which trial attributes impact participation, in either positive or negative ways, is limited. This study invites participants to record a wide range of data on their clinical trial experience, with the goal being to identify factors which persistently limit patients' ability to participate in, or complete, a trial in which they were initially interested. This data will be analyzed through a range of demographic lenses, in hopes of discovering patterns which might improve the experience of future rheumatoid arthritis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with rheumatoid arthritis
* Patient has self-identified as planning to enroll in an interventional clinical trial
* Patient is 18 years old

Exclusion Criteria:

* ECOG score of 4
* Patient is pregnant
* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients who are actively considering enrolling in an interventional clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Patient decides to enroll in clinical trial | 3 Months
Patient remains in clinical trial to completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McKinney M, Bell R, Samborski C, Attwood K, Dean G, Eakle K, Yu W, Edge S. Clinical Trial Participation: A Pilot Study of Patient-Identified Barriers. Clin J Oncol Nurs. 2021 Dec 1;25(6):647-654. doi: 10.1188/21.CJON.647-654. PMID 34800100
- [Background] Lansey DG, Hefka TA, Carducci MA, Kanarek NF. Problem Solving to Enhance Clinical Trial Participation Utilizing a Framework-Driven Approach. Clin Adv Hematol Oncol. 2020 Aug;18(8):468-476. PMID 32903246
- [Background] Michos ED, Van Spall HGC. Increasing representation and diversity in cardiovascular clinical trial populations. Nat Rev Cardiol. 2021 Aug;18(8):537-538. doi: 10.1038/s41569-021-00583-8. No abstract available. PMID 34108677

DOCUMENTS (1):
  • Informed Consent Form (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT05398471/ICF_001.pdf